CLINICAL TRIAL: NCT05444192
Title: Comparing the Effectiveness of Computer-aided-design Computer-aided-manufacture (CAD/CAM) Insoles Manufactured From Foam-box Cast vs Direct Scan on Patient Reported Outcome Measures: A Double-blinded, Randomised Controlled Trial
Brief Title: Comparing Clinical Outcomes Using Two Insole Manufacture Techniques
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: NHS Greater Glasgow and Clyde (Other)
Collaborators: University of Central Lancashire (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: GN22OR165
Record Dates: First submitted 2022-06-16; First posted 2022-07-05 (Actual); Results first posted 2025-05-23 (Actual); Last update posted 2025-05-23 (Actual); Status verified 2025-05

CONDITIONS: Foot Injury; Foot Deformity; Foot Sprain; Feet, Flat; Foot Ankle Injuries
MeSH Terms: conditions — Foot Injuries; Foot Deformities; Flatfoot

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- insoles manufactured from foam-box cast (Active Comparator): Both arms are currently standard treatment within the NHS GGC Orthotic Department. There are no experimental interventions in the study.
  Interventions: Device: CAD/CAM insoles
- insoles manufactured from direct 3D scan (Active Comparator): Both arms are currently standard treatment within the NHS GGC Orthotic Department. There are no experimental interventions in the study.
  Interventions: Device: CAD/CAM insoles

INTERVENTIONS:
Device: CAD/CAM insoles — computer-aided-design computer-aided-manufacture (CAD/CAM) insoles

SUMMARY:
The main purpose of this study is to find out if scanning the foot using a 3D scanner influences the effectiveness of custom made insoles, compared to the more traditional approach of taking a foam-box impression cast of the foot. Both of these methods are currently used as standard care in the NHS Greater Glasgow and Clyde (GGC) Orthotic Department. In this study, insoles will be manufactured either from a direct 3D scan of the foot, or from a foam-box impression cast, and a series of questionnaires will be used to measure any changes in foot pain and foot function. The results from this study will be used to develop an information resource for both patients and Orthotists which will fill gaps in our current knowledge and hopefully guide us further in providing the best possible care for future patients who require insoles.

DETAILED DESCRIPTION:
A single centre, double blinded, randomised controlled trial. Interventional, equivalence Trial design.

Participants will be asked to attend 2 face-to-face appointments for assessing and fitting of insoles, which is standard practice in the NHS GGC Orthotic Department. Each face-to-face appointment will take approximately 40 minutes. Following the fitting of the insoles, participants will be asked to participate in 3 telephone calls over 12-weeks, during which they will be asked to answer questions from two questionnaires (the "Foot Health Status Questionnaire", and the "Orthotic and Prosthetic User Survey"). Each telephone appointment will take approximately 15 minutes. Once participants receive their insoles, they will also be asked to keep a diary detailing the number of hours that they wore the insoles each day over 12-weeks. This information will be collected by the Orthotist involved with the trial during the telephone review appointments.

ELIGIBILITY:
Inclusion Criteria:

* Are aged 18 years or above
* Are referred to the NHS GGC Orthotic service requiring a new assessment for insoles
* are deemed suitable for CAD/CAM insoles as assessed by the PI or Co-I on clinical assessment
* Are able to commit to five appointments over a 16-week period (two Face-to-Face appointments, three Telephone Appointments)
* Have suitable own footwear that can accommodate a CAD/CAM insole as assessed by the PI or Co-I, and as per standard practice can wear these for 12-weeks
* Is willing to allow their General Practitioner and consultant, if appropriate, to be notified of participation in the trial.
* An adequate understanding of written and verbal information in English in order to provide informed consent and answer the study questionnaires

Exclusion Criteria:

* Scheduled elective surgery or other procedures which is likely to affect mobility during the trial.
* Scheduled steroid injection of the foot or ankle up to 3 months prior to joining the trial, or during participation in the trial
* Age <18 years
* Adult with Incapacity, under The Adults with Incapacity (Scotland) Act 2000
* Participant unable or unwilling to consent
* Medial longitudinal Arch height of the foot exceeds depth of EVA blank (35mm)
* Clinical assessment concludes that the participant requires an insole material other than EVA
* Clinical assessment concludes that the participant does not require or will be unlikely to benefit from CAD/CAM insoles.
* The participant is unable to commit to the trial conditions.
* Peripheral Neuropathy present
* Active foot ulceration present
* Participant with life expectancy of less than 6 months.
* Any other significant disease or disorder which, in the opinion of the PI or Co-I, may either put the participants at risk because of participation in the trial, or may influence the result of the trial, or the participant's ability to participate in the trial.
* Participants who have participated in another research trial involving an investigational foot orthosis in the past 12 weeks.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 114 (Actual)
Dates: Start 2022-09-29 (Actual); Primary Completion 2023-11-24 (Actual); Study Completion 2023-11-24 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Graham Chapman, Principal Investigator — University of Central Lancashire
Locations (1):
- Orthotics Department, Glasgow Royal Infirmary, Glasgow, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
Anonymised data available on request via email to the corresponding author
Supporting Information: Study Protocol, SAP, ICF, Analytic Code
Time Frame: Data is available after publication
Access Criteria: For academic and research purposes

REFERENCES:
- [Derived] Barr L, Richards J, Dickson C, Tawse J, Munro N, Scott H, Holland A, Chapman GJ. To scan or not to scan? Comparing the effectiveness and cost differential of insoles manufactured from foam-box casts versus direct scans in treating musculoskeletal conditions of the foot and ankle: a double-blinded, randomised controlled trial. BMC Musculoskelet Disord. 2025 Mar 22;26(1):282. doi: 10.1186/s12891-025-08513-2. PMID 40121418
- [Derived] Barr L, Richards J, Chapman GJ. Comparing the effectiveness of computer-aided design/computer-aided manufacturing (CAD/CAM) of insoles manufactured from foam box cast versus direct scans on patient-reported outcome measures: a protocol for a double-blinded, randomised controlled trial. BMJ Open. 2024 Apr 2;14(4):e078240. doi: 10.1136/bmjopen-2023-078240. PMID 38569685

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Assessed for eligibility (n=118) Excluded (n=4)
  * Already has suitable insoles (n=2)
  * Not suitable for treatment with insoles (n=1)
  * Declined to participate (n=1)
Period: Overall Study
Arm/Group | Insoles Manufactured From Foam-box Cast | Insoles Manufactured From Direct 3D Scan
Started | 57 | 57
Completed | 56 | 57
Not Completed | 1 | 0
Not completed — Lost to Follow-up | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Insoles Manufactured From Foam-box Cast | Insoles Manufactured From Direct 3D Scan | Total
Number analyzed (Participants) | 57 | 57 | 114
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 50.0 [32.0 to 61.0] | 50.0 [34.0 to 59.0] | 50.0 [33.0 to 60.0]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 41 | 41 | 82
  Male | 16 | 16 | 32
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Ethnicity: White | 56 | 56 | 112
  Ethnicity: Other (mixed) | 0 | 1 | 1
  Ethnicity: African | 1 | 0 | 1
Area of primary musculoskeletal pathology [Count of Participants; unit: Participants] — A review of all relevant medical history from the participant's medical record was undertaken to determine primary pathology, in conjunction with a physical examination of the foot and ankle, including the following standard biomechanical tests
  1. Foot Posture Index
  2. Jacks test for Functional Hallux Limitus
  3. Palpation technique for Subtalar Joint Axis Location
  4. Passive assessment of ankle dorsiflexion stiffness by 'position of first detectable resistance
  5. Supination resistance test
  6. Visual gait analysis
  Participants
    Ankle | 21 | 24 | 45
    First ray | 3 | 10 | 13
    Forefoot | 17 | 10 | 27
    Lower leg | 0 | 1 | 1
    Midfoot | 4 | 1 | 5
    Plantar heel / plantar fascia | 12 | 11 | 23

OUTCOME MEASURES:

1. Primary Outcome: Foot Health Status Questionnaire (FHSQ) - Pain Sub-domain
Description: To compare the changes in pain in two groups of participants fitted with custom CAD/CAM insoles manufactured using different foot shape capture methods. Units on a scale. Minimum score is 0, maximum score is 100. Higher scores represent better outcomes.
Time Frame: Measured 4 times throughout the 12-week period that the participant is wearing the insoles: Baseline immediately after receiving intervention (insoles). 4 weeks after intervention. 8 weeks after intervention. And 12 weeks after intervention
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | Insoles Manufactured From Foam-box Cast | Insoles Manufactured From Direct 3D Scan
Number analyzed (Participants) | 56 | 57
units on a scale
  12 weeks following intervention | 78.13 [53.75 to 92.97] | 78.75 [53.75 to 93.75]
  8 weeks following intervention | 72.50 [49.53 to 84.38] | 78.13 [54.06 to 85.00]
  4 weeks following intervention | 72.50 [57.19 to 84.38] | 78.13 [48.13 to 84.38]
  Baseline | 48.13 [29.38 to 71.88] | 53.75 [27.19 to 72.50]

2. Secondary Outcome: Foot Health Status Questionnaire (FHSQ) - Function Sub-domain
Description: To compare the changes in foot function in two groups of participants fitted with custom CAD/CAM insoles manufactured using different foot shape capture methods. Units on a scale. Minimum score is 0, maximum score is 100. Higher scores represent better outcomes.
Time Frame: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | Insoles Manufactured From Foam-box Cast | Insoles Manufactured From Direct 3D Scan
Number analyzed (Participants) | 56 | 57
units on a scale
  12 weeks following intervention | 87.50 [68.75 to 100.00] | 93.75 [65.63 to 100.0]
  8 weeks following intervention | 75.00 [51.56 to 93.75] | 93.75 [59.38 to 100.00]
  4 weeks following intervention | 87.50 [57.81 to 93.75] | 87.50 [62.50 to 100.00]
  Baseline | 68.75 [43.75 to 87.50] | 62.50 [37.50 to 90.63]

3. Secondary Outcome: Foot Health Status Questionnaire - Foot Health Sub-domain
Description: To compare the changes in foot health in two groups of participants fitted with custom CAD/CAM insoles manufactured using different foot shape capture methods. Units on a scale. Minimum score is 0, maximum score is 100. Higher scores represent better outcomes.
Time Frame: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | Insoles Manufactured From Foam-box Cast | Insoles Manufactured From Direct 3D Scan
Number analyzed (Participants) | 56 | 57
units on a scale
  12 weeks following intervention | 60.00 [25.00 to 81.88] | 72.50 [25.00 to 85.00]
  8 weeks following intervention | 46.25 [25.00 to 69.38] | 72.50 [25.00 to 85.00]
  4 weeks following intervention | 42.50 [25.00 to 72.50] | 60.00 [25.00 to 85.00]
  Baseline | 25.00 [0.00 to 60.00] | 42.50 [0.00 to 72.50]

4. Secondary Outcome: Orthotic and Prosthetic User Survey9-12 (Satisfaction With Device Survey)
Description: To compare the patient satisfaction in two groups of participants fitted with custom CAD/CAM insoles manufactured using different foot shape capture methods. Units on a scale. Minimum score is 0, maximum score is 100. Higher scores represent better outcomes.
Time Frame: Measured 12 weeks after being fitted with insoles
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Insoles Manufactured From Foam-box Cast | Insoles Manufactured From Direct 3D Scan
Number analyzed (Participants) | 55 | 57
units on a scale | 69.48 [64.59 to 74.36] | 76.35 [71.84 to 80.86]

5. Secondary Outcome: Differential Cost Analysis
Description: A differential cost analysis was undertaken. This involved calculating the total cost for each participant using a calculation of transit costs, staff time, and physical resources for each participant throughout their time in the trial.
Time Frame: Costs were calculated per participant from baseline until their completion of the trial at week 12.
Measure: Mean (95% Confidence Interval); unit: cost in pounds and pence per participant
Arm/Group | Insoles Manufactured From Foam-box Cast | Insoles Manufactured From Direct 3D Scan
Number analyzed (Participants) | 57 | 57
cost in pounds and pence per participant | 55.46 [51.28 to 60.36] | 44.94 [39.98 to 48.12]

6. Other Pre Specified Outcome: Tertiary Outcome Measure - Hours of Insole Wear Time Per Day
Description: Patients will keep a diary of daily wear time in hours, in accordance with prior publications on measuring Orthotic Adherence. The minimum threshold for adherence is >21 hours per week
Time Frame: Measured from baseline until completion of the trial at week 12
Measure: Mean (95% Confidence Interval); unit: Hours
Arm/Group | Insoles Manufactured From Foam-box Cast | Insoles Manufactured From Direct 3D Scan
Number analyzed (Participants) | 56 | 57
Hours | 5.08 [4.66 to 5.50] | 6.09 [5.68 to 6.51]

7. Other Pre Specified Outcome: Tertiary Outcome Measure - Dropout Rate
Description: Dropout rate = n dropout at end of trial
Time Frame: Measured from baseline to completion of the trial at 12 weeks, for each participant
Measure: Count of Participants; unit: Participants
Arm/Group | Insoles Manufactured From Foam-box Cast | Insoles Manufactured From Direct 3D Scan
Number analyzed (Participants) | 57 | 57
Participants | 2 | 0

ADVERSE EVENTS:
Time Frame: 14 months
Arm/Group | Insoles Manufactured From Foam-box Cast | Insoles Manufactured From Direct 3D Scan
All-Cause Mortality (participants affected / at risk) | 0/57 | 0/57
Serious Adverse Events (participants affected / at risk) | 0/57 | 0/57
Other Adverse Events (participants affected / at risk) | 7/57 | 2/57
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Insoles Manufactured From Foam-box Cast (N=57) | Insoles Manufactured From Direct 3D Scan (N=57)
Advenrse event (Skin and subcutaneous tissue disorders) | 7 (7) | 2 (2) — Discomfort in the arch area of the foot (n=7), the lateral midfoot (n=1) and the forefoot (n=1).

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2022-09-08): https://cdn.clinicaltrials.gov/large-docs/92/NCT05444192/Prot_SAP_000.pdf
  • Informed Consent Form (2022-09-08): https://cdn.clinicaltrials.gov/large-docs/92/NCT05444192/ICF_001.pdf